CLINICAL TRIAL: NCT01414426
Title: Randomized Placebo- Controlled Pilot Study of ZD6474 as a Chemopreventive Agent for Premalignant Lesions of the Head and Neck
Brief Title: Vandetanib in Preventing Head and Neck Cancer in Patients With Precancerous Head and Neck Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11-0265; NCI-2011-01246 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Lip and Oral Cavity Squamous Cell Carcinoma; Oral Cavity Verrucous Carcinoma; Precancerous Condition
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia; Squamous Cell Carcinoma of Head and Neck; Precancerous Conditions | interventions — vandetanib; Immunohistochemistry; Biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (chemoprevention) (Experimental): Patients receive vandetanib PO QD for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vandetanib; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: biopsy; Other: pharmacological study
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: biopsy; Other: pharmacological study

INTERVENTIONS:
Drug: vandetanib — Given PO
  Other Names: AZD6474; ZD6474
  Arms: Arm I (chemoprevention)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: laboratory biomarker analysis — Correlative studies
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This randomized phase II trial studies how well vandetanib works in preventing head and neck cancer in patients with precancerous head and neck lesions. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of vandetanib may keep cancer from forming in patients with premalignant lesions

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effect of ZD6474 (vandetanib) compared to placebo on microvessel density (MVD) from baseline to 3 months in patients at risk for oral squamous cell carcinoma (OSCC) with preneoplastic lesions.

SECONDARY OBJECTIVES:

I. Change in MVD over 6 months. II. Change in putative targets of ZD6474: tissues will be analyzed by immunohistochemistry (IHC) for phosphorylated epidermal growth factor receptor (pEGFR), EGFR, phosphorylated-vascular endothelial growth factor receptor 2 (pVEGFR2), VEGFR2.

III. Change in proliferative index as measured by Ki-67 IHC. IV. Safety, tolerability, and adherence to ZD6474 for 6 months in patients at risk for OSCC.

TERTIARY OBJECTIVES:

I. Compare OSCC incidence in both study arms (ZD6474 and placebo).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive vandetanib orally (PO) once daily (QD) for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO QD for 6 months. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 9 and 12 months and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological confirmation of oral cavity dysplasia and one of three additional criteria:
* Prior history of OSCC
* Loss of heterozygosity (LOH) at 3p or 9p
* Expression by immunohistochemistry (IHC) of budding uninhibited by benzimidazoles 3 (BUB3)/sex determining region Y (SOX4)
* Provision of informed consent
* Females of child bearing age must have a negative serum pregnancy test within 7 days of first dose of study drug
* Patients must not have been taking steroids or are on a stable dose of steroids for at least 14 days before enrollment
* Patients must have a Karnofsky Performance Score of 70% or above

Exclusion Criteria:

* History of malignancy within the last 5 years other than squamous cell carcinoma of the head and neck (SCCHN) and superficial non-melanoma skin cancer; patients with a history of SCCHN must be free of active carcinoma
* Currently receiving treatment for any malignancy
* Serum bilirubin > 1.5x the upper limit of reference range (ULRR)
* Creatinine clearance =< 30 mL/minute (calculated by Cockcroft-Gault formula)
* Potassium, < 4.0 mmol/L despite supplementation; or above the Common Terminology Criteria for Adverse Events (CTCAE) grade 1 upper limit
* Magnesium below the normal range despite supplementation, or above the CTCAE grade 1 upper limit
* Serum calcium above the CTCAE grade 1 upper limit; in cases where the serum calcium is below the normal range, 2 options would be available: 1) the calcium adjusted for albumin is to be obtained and substituted for the measured serum value; exclusion is to then be based on the adjusted for albumin values falling below the normal limit; 2) Determine the ionized calcium levels; if these ionized calcium levels are out of normal range despite supplementation, then the patient must be excluded
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × ULRR
* Alkaline phosphatase (ALP) > 2.5 x ULRR
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Clinically significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome [SVC], New York Heart Association [NYHA] classification of heart disease > 2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia
* History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation), which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia; atrial fibrillation, controlled on medication is not excluded
* QTc prolongation with other medications that required discontinuation of that medication
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age
* Presence of left bundle branch block (LBBB)
* QTc with Bazett's correction that is unmeasurable or ≥450 msec on screening electrocardiogram (ECG); (Note: If a subject has a QTc interval >= 450 msec on screening ECG, the screen ECG may be repeated twice [at least 24 hours apart]; the average QTc from the three screening ECGs must be < 450 msec in order for the subject to be eligible for the study)
* Any concurrent medication with a known risk of inducing Torsades de Pointes, that in the investigator's opinion cannot be discontinued
* Concomitant medications that are potent inducers (rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital and St. John's Wort) of Cytochrome P450 3A4 (CYP3A4) function
* Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm mercury (Hg) or diastolic blood pressure greater than 100 mm Hg)
* Currently active diarrhea that may affect the ability of the patient to absorb the ZD6474 or tolerate diarrhea
* Women who are currently pregnant or breast-feeding
* Receipt of any investigational agents within 30 days prior to commencing study treatment
* Previous enrollment or randomization of treatment in the present study
* Major surgery within 4 weeks or incompletely healed surgical incision before starting study therapy
* Involvement in the planning and conduct of the study (applies to both Astra Zeneca staff and staff at the study site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Chemoprevention) | Arm II (Placebo)
Started | 10 | 10
Completed | 9 | 8
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemoprevention) | Arm II (Placebo) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.0) | 49.0 (15.0) | 54.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 1 | 6 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Comparison Between Treatment Groups of the Within-patient Change in MVD Score Following Treatment Initiation
Description: A Wilcoxon ranksum test may be used if the normality assumption is not satisfied. Alternatively, change in MVD may be transformed (e.g. log-transformation) to satisfy the normality assumption. Additional analyses will include linear regression models with treatment effect and other prognostic factors as covariates.
Time Frame: Baseline to 3 months
Population: The outcome measure microvessel density was not collected on any subjects
Arm/Group | Arm I (Chemoprevention) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events rate shows the total number of subjects with an AE.
Time Frame: Weekly during treatment, up to week 24
Measure: Number; unit: participants
Arm/Group | Arm I (Chemoprevention) | Arm II (Placebo)
Number analyzed (Participants) | 10 | 10
participants
  Week 1 | 3 | 6
  Week 2 | 4 | 3
  Week 3 | 0 | 1
  Week 4 | 2 | 0
  Week 5 | 5 | 5
  Week 6 | 0 | 2
  Week 7 | 0 | 0
  Week 8 | 0 | 0
  Week 9 | 7 | 2
  Week 10 | 0 | 1
  Week 11 | 0 | 0
  Week 12 | 0 | 0
  Week 13 | 3 | 0
  Week 14 | 0 | 0
  Week 15 | 0 | 0
  Week 16 | 0 | 1
  Week 17 | 2 | 1
  Week 18 | 0 | 2
  Week 19 | 0 | 0
  Week 20 | 0 | 1
  Week 21 | 1 | 0
  Week 22 | 0 | 1
  Week 23 | 2 | 0
  Week 24 | 0 | 0
  Week 25 | 2 | 0

3. Secondary Outcome: Number of Participants Who Adhered to Treatment
Description: Number of participants who Adhered to Treatment
Time Frame: Over 6 months
Measure: Number; unit: participants
Arm/Group | Arm I (Chemoprevention) | Arm II (Placebo)
Number analyzed (Participants) | 10 | 10
participants | 4 | 5

4. Secondary Outcome: Development of Oral and Other Cancers
Description: Number of patients with new cancer
Time Frame: At 6, 9, and 12 months and then ever 6 months for 2 years
Measure: Number; unit: participants
Arm/Group | Arm I (Chemoprevention) | Arm II (Placebo)
Number analyzed (Participants) | 10 | 10
participants
  6 months | 1 | 0
  9 months | 0 | 0
  12 months | 0 | 0
  18 Months | 0 | 0
  24 Months | 0 | 0

5. Secondary Outcome: Biologic Effect of EGFR and VEGFR2 Inhibition
Description: Effect of treatment on EGFR and VEGFR2 inhibition
Time Frame: Baseline and 3 and 6 months
Population: Outcome measure was not collected.
Arm/Group | Arm I (Chemoprevention) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 180 days
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Arm/Group | Arm I (Chemoprevention) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Chemoprevention) (N=10) | Arm II (Placebo) (N=10)
Gastrointestinal (Gastrointestinal disorders) | 6 (8) | 4 (6)
General (Product Issues) | 4 (5) | 3 (5)
Infections (Infections and infestations) | 1 (1) | 1 (1)
Metabolic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Nervous System (Nervous system disorders) | 2 (3) | 1 (1)
Psychiatric (Psychiatric disorders) | 0 (0) | 2 (2)
Renal (Renal and urinary disorders) | 1 (1) | 0 (0)
Skin (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (5)
Vascular (Vascular disorders) | 2 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT01414426/Prot_SAP_000.pdf